CLINICAL TRIAL: NCT04714619
Title: CB-103 Plus NSAI In Luminal Advanced Breast Cancer: CAILA Study
Brief Title: CB-103 Plus NSAI In Luminal Advanced Breast Cancer
Acronym: CAILA
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: MedSIR (Other)
Collaborators: Cellestia Biotech AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MedOPP319
Record Dates: First submitted 2020-12-02; First posted 2021-01-19 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2022-06

CONDITIONS: Advanced Breast Cancer
MeSH Terms: interventions — Letrozole; Anastrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- CB-103 + NSAI therapy (Experimental): Hormone Receptor (HR)-positive and HER2-negative advanced breast cancer, including metastatic (ABC).Approximately 80 patients
  Interventions: Drug: CB-103

INTERVENTIONS:
Drug: CB-103 — Patients will receive CB-103 capsules orally (QD) in combination with NSAI therapy (letrozole or anastrozole, continuing prior therapy) also orally once daily, and based on a 28-day treatment cycle.
  A run-in phase for safety and tolerability of CB-103 in combination with anastrozole or letrozole will be conducted as an initial step of the phase II trial to confirm the safe dose of CB-103 in combination with NSAI given at standard dose.
  Patients will receive treatment until disease progression (as defined by RECIST v.1.1), symptomatic deterioration, unacceptable toxicity, death, consent withdrawal or study termination, whichever occurs first.
  Other Names: Letrozole; Anastrozole

SUMMARY:
Multicenter, single-arm, open label, phase II clinical trial with safety run-in to evaluate the safety, tolerability, pharmacokinetics and efficacy of CB-103 in combination with a non-steroidal aromatase inhibitor (NSAI), anastrozole or letrozole, in Hormone Receptor-positive and Human Epidermal Growth Factor Receptor 2 (HER2)-negative advanced breast cancer patients who have achieved clinical benefit during prior NSAI-based treatment.

DETAILED DESCRIPTION:
This is a ulticenter, single arm, open-label, Phase II clinical trial to evaluate the safety, tolerability, pharmacokinetics, and efficacy of CB-103 in combination with a non-steroidal aromatase inhibitor (NSAI), anastrozole or letrozole, in Hormone Receptor-positive and Human Epidermal Growth Factor Receptor 2 (HER2)-negative advanced breast cancer patients who have achieved clinical benefit during prior NSAI-based treatment.

Eligible patients include pre- and post-menopausal women age ≥ 18 years with HR-positive and HER2-negative unresectable advanced breast cancer (ABC, including metastatic), having achieved at least clinical benefit upon treatment with prior NSAI. Evidence of measurable or evaluable disease, as per RECIST (Response Evaluation Criteria In Solid Tumors) v.1.1, with a tumor lesion amenable to biopsy. Pre-menopausal women must be under treatment with luteinizing hormone-releasing hormone (LHRH) analogues. Patients are not eligible if they are candidates for a local treatment with a curative intention

The primary objective is to assess the efficacy, defined as progression-free survival (PFS), of CB-103 in combination with NSAI therapy (anastrozole or letrozole) in women with HR-positive, HER2-negative, unresectable ABC with evidence of Notch signaling pathway activation and with progressive disease after clinical benefit while on prior NSAI-containing regimen.

Approx 80 patients are expected to be recruited

ELIGIBILITY:
Inclusion Criteria:

Patients must meet ALL of the following inclusion criteria to be eligible for enrolment into the study:

1. Signed the informed consent form (ICF) prior to any study-related activities.
2. Female patients ≥ 18 years of age at time of ICF signature.
3. Pre- or peri-menopausal women being treated with a LHRH analogue for at least 28 days prior to study entry (if shorter, post-menopausal levels of serum estradiol/Follicle-stimulating hormone [FSH] must be confirmed analytically), or post-menopausal women as defined by any of the following criteria:

   1. Age ≥60 years;
   2. Age <60 years and cessation of regular menses for at least 12 consecutive months with no alternative pathological or physiological cause; and serum estradiol and/or FSH level within the laboratory's reference range for postmenopausal females;
   3. Documented bilateral oophorectomy.
4. Eastern Cooperative Oncology Group (ECOG) performance status lower or equal to 1.
5. Life expectancy greater or equal to 6 months.
6. Locally advanced or metastatic breast cancer not amenable to treatment with curative intend.
7. Histologically confirmed ER-positive and/or PgR-positive (with ≥10% positive stained cells according to National Comprehensive Cancer Network and American Society of Clinical Oncology guidelines) and HER2-negative (0-1+ by immunohistochemistry [IHC] or 2+ and negative by in situ hybridization [ISH] test) breast cancer based on local testing on the most recent analyzed biopsy.
8. Patients with radiological evidence (as per RECIST v.1.1) of disease progression on the immediate prior line of treatment containing a non-steroidal aromatase inhibitor (NSAI) (anastrozole-letrozole). Patients must meet at least one of the following conditions:

   1. On adjuvant endocrine therapy for ≥ 24 months and relapsing within 12 months after CDK4/6 inhibitor treatment completion following the adjuvant setting.
   2. Progression to an NSAI in the advanced setting (with or without a CDK4/6 inhibitor) after obtaining clinical benefit (stable disease for ≥ 6 months, CR or PR) Note: Last dose of NSAI (anastrozole or letrozole) of the prior ET must have been received within the 28 days before starting study treatment.
9. At least 1 and no more than 3 prior lines of endocrine therapy for ABC, including the treatment received at the time of study entry. ET might have been combined with targeted agents such as everolimus, PI3K inhibitors, CDK4/6 inhibitors, etc.
10. Evidence of measurable or non-measurable disease according to RECIST v.1.1. Patients with only bone lesions are not eligible.

    Note: Previously irradiated lesions can be considered as measurable disease only if disease progression has been unequivocally documented at that site since radiation.
11. Willingness and ability to provide tumor biopsy at study entry (available tumor tissue sample from a fresh pre-treatment core or excisional biopsies).

    In the case of biopsable lesions that can be safely accessed, the patient should also consent to a biopsy at the time of start of Cycle 2 (C2D1 ± 3 days), unless investigator considers there are any medical concerns. These cases will be discussed with Sponsor medical monitor on a case by case basis.

    At disease progression, a tumor biopsy will be requested if there are accessible lesions.

    If available, patients will be asked to provide archived primary or metastatic tumor specimen, but consent will not be limiting for enrolment.
12. Patients agree to collection of blood samples for molecular analysis.
13. Adequate hematological and organ function within 14 days before the first CB 103 dose:

    a. Hematological (without platelet transfusion or granulocyte colony-stimulating factor [G-CSF] support within 14 days before first CB 103 dose): i. White blood cell (WBC) count > 3.0 x 109/L; ii. Absolute neutrophil count (ANC) > 1.5 x 109/L; iii. Platelet count > 75.0 x109/L; iv. Hemoglobin > 10.0 g/dL. b. Hepatic: i. Serum albumin ≥ 3 g/dL; ii. Total bilirubin ≤ 1.5 times the upper limit of normal (× ULN) (< 3 x ULN in the case of Gilbert's disease); iii. Aspartate transaminase (AST), and alanine transaminase (ALT) ≤ 3.0 times × ULN (in the case of liver metastases ≤ 5 × ULN); iv. Alkaline phosphatase (ALP) ≤ 2.5 times × ULN (≤ 5 × ULN in the case of liver and/or bone metastases ≤ 5 × ULN).

    c. Renal: i. Serum creatinine ≤ 1.5 x ULN or creatinine clearance ≥ 30 mL/min based on Cockcroft-Gault glomerular filtration rate estimation.

    d. Coagulation: i. Partial thromboplastin time (PTT) ≤ 1.5 x ULN (or activated Partial Thromboplastin Time [aPTT]) and international normalized ratio (INR) ≤ 1.5 times × ULN.
14. Patients who are willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.
15. Women of childbearing potential must have a negative serum pregnancy test within 7 days before start of study treatment. These women must agree to remain abstinent (refrain from heterosexual intercourse) or use highly effective contraceptive methods, or two effective contraceptive methods (as defined in the protocol) during the treatment period and for at least 90 days after the last dose of CB 103, and agreement to refrain from donating eggs during this same period.
16. Resolution of all acute toxic effects of prior anti-cancer therapy to Grade ≤ 1 as determined by the National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE) v.5.0 (except for alopecia or other toxicities, such as myelosuppression, not violating other inclusion criteria and not considered a safety risk for the patient at investigator's discretion).

Exclusion Criteria:

Patients will be excluded from the study if they meet ANY of the following criteria:

1. Prior chemotherapy and/or Notch signaling inhibitors treatment (e.g., gamma-secretase inhibitors) in the metastatic setting.
2. Treatment with any approved or investigational cancer therapy between the end of NSAI treatment and study entry.
3. Rapidly or symptomatic progressive visceral disease or any disease burden that contraindicates continuing ET according to Investigator's judgement.
4. Known active uncontrolled or symptomatic central nervous system (CNS) metastases, carcinomatous meningitis, or leptomeningeal disease as indicated by clinical symptoms, cerebral edema, and/or progressive growth. Patients with a history of CNS metastases or cord compression are eligible if they have been definitively treated (e.g., radiotherapy, stereotactic surgery) and are neurologically stable off anticonvulsants and steroids for at least 4 weeks before start of treatment.
5. Receiving any of following concomitant medications that cannot be discontinued during the study treatment duration (see Section 6.9 and 6.10 for more details):

   1. Drugs which prolong QT interval, either with a known or a conditional/ possible risk to induce Torsades de Pointes (listed in Appendix 3).
   2. Coumarin-type anticoagulants (such as warfarin) within one week prior first CB 103 dose. Low molecular weight heparin and direct oral anticoagulants are permitted.
6. Current or prior malignancy within 5 years prior to study enrolment, except non-melanoma skin cancer, or carcinoma in situ of the uterine cervix. Patients with other cancers considered to have a low risk of recurrence might be included after approval by the Medical Monitor.
7. Radiotherapy or limited-field palliative radiotherapy within 7 days prior to enrolment or patients not having recovered from radiotherapy-related toxicities to baseline or Grade ≤ 1 and/or from whom ≥ 25% of the bone marrow has been previously irradiated.
8. Inability to swallow capsules or tablets.
9. Impairment of gastrointestinal function or presence of gastrointestinal disease that may significantly alter the absorption of CB-103.
10. Impaired cardiac function or clinically significant cardiac disease, including any of the following:

    1. Clinically significant cardiac disease including congestive heart failure (New York Heart Association [NYHA] class III or IV), arrhythmia or conduction abnormality requiring medication, or cardiomyopathy
    2. Clinically uncontrolled hypertension (systolic blood pressure > 160 or diastolic blood pressure >110 mmHg).
    3. Complete left bundle branch block.
    4. Right bundle branch block and left anterior hemiblock
    5. Mandatory use of a cardiac pacemaker.
    6. Congenital long QT syndrome.
    7. History or presence of sustained or symptomatic ventricular tachyarrhythmia.
    8. Presence of atrial fibrillation.
    9. Clinically significant resting bradycardia (< 50 bpm).
    10. Corrected QT interval using Fridericia formula (QTcF) > 470 ms at the Screening ECG.
    11. QRS ≥ 110 ms.
    12. History of symptomatic congestive heart failure.
    13. Left ventricular ejection fraction (LVEF) < 50%. History of absolute decrease in LVEF of ≥ 15 absolute percentage points, or ≥ 10 absolute percentage points and crossing from > lower limits of normal (LLN) to < LLN on anticancer therapy, even if asymptomatic.
    14. Angina pectoris ≤ 6 months prior to first CB 103 dose.
    15. Acute myocardial infarction (MI) ≤ 6 months prior to starting study drug.
11. General conditions or other clinically significant diseases, including any one of the following:

    1. Hemorrhagic, embolic, or thrombotic stroke within 6 months prior to the first CB-103 dose
    2. Prior allogeneic bone marrow/hematopoietic stem cell transplant
    3. Prior autologous hematopoietic stem cell transplant for breast cancer (for other indications within ≤ 6 months prior first CB 103 dose.
    4. Known infection with human immunodeficiency virus (HIV) or hepatitis B or C requiring treatment.
    5. Any active infection requiring the use of parenteral anti-microbial agents or that is > Grade 2.
    6. Non-malignant interstitial lung disease or pneumonitis.
    7. Dyspnea of any cause requiring supplemental oxygen therapy and dyspnea at rest due to complications of advanced malignancy and co-morbidities.
    8. Significant traumatic injury or major surgery (i.e., opening of a body cavity, e.g., thoracotomy, laparotomy, laparoscopic organ resection) or major orthopedic procedures (e.g. joint replacement, open reduction and internal fixation) within 14 days prior first CB-103 dose.
    9. Other concurrent severe and/or uncontrolled medical conditions (e.g. uncontrolled diabetes, active or uncontrolled infection) that could cause unacceptable safety risks or compromise compliance with the protocol.
12. Hypersensitivity to CB-103 or any of its excipients.
13. Pregnant or breast-feeding patients.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2021-05-06 (Actual); Primary Completion 2021-09-02 (Actual); Study Completion 2022-04-26 (Actual)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | from treatment initiation until objective tumor progression or death
  PFS, defined as the time from treatment initiation until objective tumor progression or death from any cause, whichever occurs first, as per Investigator assessment by Response Evaluation Criteria in Solid Tumors (RECIST) version (v) 1.1 in the subgroup of patients with evidence of Notch signaling pathway activation.We hypothesize that excluding a median PFS of 2 months while targeting an improvement of the median PFS greater than or equal to 4 months (hr = 0.50) in patients with evidence of Notch pathway activation is an optimal approach to evaluate the clinical activity of the CB-103 plus NSAI (anastrozole or letrozole) combination.

SECONDARY OUTCOMES:
Safety and tolerability of CB-103 in combination with NSAI (anastrozole or letrozole) | from baseline until end of study.All patients must be followed for AEs and SAEs for 28 days following the last dose of study drug.
  Incidence and severity of AEs and SAEs according to the NCI-CTCAE v.5.0, including dose reductions, delays, and treatment discontinuations.
Efficacy in terms of PFS of CB-103 in combination with NSAI in all patients and in sub.groups | from treatment initiation until objective tumor progression or death (at least 4months)
  PFS, defined as the time from treatment initiation until objective tumor progression or death from any cause, whichever occurs first, as per Investigator assessment by RECIST v.1.1 in all patients and in patients without evidence of Notch signaling pathway activation.
Overall response rate (ORR) | from baseline until end of study (will occur when all patients have discontinued treatment or 12 month after the last patient was enrolled on the study plus the safety follow up window of 28 days after last dose of study treatment in the last patient)
  ORR, defined as the proportion of patients with complete response (CR) or partial response (PR), as per Investigator assessment using RECIST v.1.1., in patients with and without evidence of Notch signalling pathway activation.
Clinical benefit rate (CBR) | 24 weeks
  CBR at 24 weeks, defined as the proportion of patients who obtain an objective response (CR or PR), or stable disease for at least 24 weeks, as per Investigator assessment using RECIST v.1.1., in patients with or without evidence of Notch signaling pathway activation.
Clinical benefit rate (CBR) | 12 weeks
  CBR at 12 weeks, defined as the proportion of patients who obtain an objective response (CR or PR), or stable disease for at least 12 weeks, as per Investigator assessment using RECIST v.1.1., in patients with or without evidence of Notch signaling pathway activation.
Time to tumor response (TTR) | from treatment initiation to time of the first objective tumor response up to 12 months
  TTR, defined as the time from treatment initiation to time of the first objective tumor response (tumor shrinkage of ≥ 30%) in patients who achieved a CR or PR, as per Investigator assessment using RECIST v.1.1., in patients with or without evidence of Notch signaling pathway activation.
Duration of response (DoR) | from the first occurrence of a documented objective response to disease progression or death, up to 12 months
  DoR, defined as the time from the first occurrence of a documented objective response to disease progression or death from any cause, whichever occurs first, as per Investigator assessment using RECIST v.1.1., in patients with or without evidence of Notch signaling pathway activation.
Overall survival (OS) | from baseline until end of study
  OS, defined as the time from treatment initiation to death from any cause, in patients with or without evidence of Notch signaling pathway activation.
Maximum tumor shrinkage (MTS) | from baseline until end of study (will occur when all patients have discontinued treatment or 12 month after the last patient was enrolled on the study plus the safety follow up window of 28 days after last dose of study treatment in the last patient)
  MTS from baseline in the size of target tumor lesions, defined as the biggest decrease, or smallest increase if no decrease observed, as per Investigator assessment using RECIST v.1.1.
Pharmacokinetics (PK), in terms of Cmax | from baseline until end of treatment, an average of 12 months
  Plasma PK parameters (Cmax) of CB-103, anastrozole and letrozole.
PK, in terms of AUC | from baseline until end of treatment, an average of 12 months
  Plasma PK parameters (Area under the plasma concentration versus time curve (AUC of CB-103, anastrozole and letrozole.
PK in terms of Vd/F | from baseline until end of treatment, an average of 12 months
  Plasma PK parameters (Vd/F ) of CB-103, anastrozole and letrozole.
PK in terms of CL/F | from baseline until end of treatment, an average of 12 months
  Plasma PK parameters (CL/F ) of CB-103, anastrozole and letrozole.
Pharmacokinetics (PK), in terms of Tmax | from baseline until end of treatment, an average of 12 months
  Plasma PK parameters Tmax of CB-103, anastrozole and letrozole.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Llombart-Cussac, Principal Investigator — Arnau de Vilanova Hospital, Valencia (Spain)
Locations (2):
- Spain (2):
  - Complejo Hospitalario de Jaen, Jaén
  - Hospital Sant Joan de Reus, Reus

IPD SHARING:
Plan to Share IPD: No